CLINICAL TRIAL: NCT07066943
Title: A Hybrid Type 3 Effectiveness-implementation Trial of an Online Psychotherapy Program for Mental Health Prevention Among Healthcare Professionals in the Andalusian Health System
Brief Title: Implementing Online Mental Health Program
Acronym: IM-MIND-SAS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud (Other)
Collaborators: Hospital Miguel Servet (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RHJ-0043-2024
Record Dates: First submitted 2025-07-04; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Stress; Healthcare Workers; Mindfulness; Prevention Intervention
Keywords: Third-wave psychotherapies; mindfulness; healthcare workers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MINDxYOU (Experimental): The online program MINDxYOU is based on the principles of 'third wave' psychotherapies, such as the promotion of wellbeing through the practice of mindfulness, compassion, acceptance, and spirituality and the estimated time for completing the whole program is 8 weeks
  Interventions: Behavioral: MINDxYOU

INTERVENTIONS:
Behavioral: MINDxYOU — The online program MINDxYOU is based on the principles of 'third wave' psychotherapies and it is an online program particularly addressed at healthcare providers which will both monitor and support the individual's mental health. The program is self-administered and will be delivered via the Internet and available via smartphone, tablet, and personal computer.

SUMMARY:
This study evaluates the feasibility, acceptability, and sustainability of MINDxYOU, a self-guided online psychotherapy program designed to reduce stress and improve the mental well-being of healthcare professionals in the Andalusian public health system. The trial uses a hybrid type 3 effectiveness-implementation design, combining the evaluation of implementation outcomes with observation of clinical effects on stress, anxiety, and depression. The intervention includes mindfulness, compassion, and acceptance-based practices delivered in four online modules over eight weeks. The study will be conducted in two phases: an initial hospital-based pilot and a broader rollout across primary care and hospital centers. Results will help identify how digital mental health interventions can be integrated into routine healthcare settings to support professionals working under high stress.

DETAILED DESCRIPTION:
Healthcare professionals are at risk of developing mental health disorders due to the high levels of stress they experience. Therefore, it is essential to provide evidence-based psychotherapeutic interventions aimed at reducing their stress and improving their well-being. This study presents a type III hybrid effectiveness-implementation trial that evaluates the feasibility, acceptability, and sustainability of MINDxYOU, an online psychotherapy program designed for healthcare workers. In response to the growing demand for accessible and effective psychological interventions for this population, the study aims to test an implementation strategy that facilitates the integration of an evidence-based intervention into routine clinical practice.

The current research uses a type III hybrid design that focuses on evaluating implementation strategies in real-world settings, assessing how the intervention is implemented while simultaneously collecting data on its clinical effectiveness. The study will be conducted in two phases. Phase 1 will consist of a pilot in a hospital setting, and Phase 2 will extend the implementation to the Andalusian Health Service (SAS). Participants will include healthcare professionals who provide direct patient care in hospitals or primary care centers. The implementation study will analyze feasibility, acceptability, and sustainability.

The study will involve health and social care centers, including hospitals and primary care units. The primary outcomes will be implementation-related metrics, while clinical outcomes associated with the intervention will be examined as secondary outcomes.

This implementation study will be useful in establishing a framework for addressing barriers and promoting facilitators that affect the feasibility, acceptability, and sustainability of online interventions. The ultimate goal is to help close the gap between research and clinical practice, which would contribute to reducing the high levels of stress experienced by healthcare professionals.

ELIGIBILITY:
Inclusion Criteria:

1. Being a current healthcare professional.
2. Age between 18 and 70 years.
3. Ability to understand Spanish.
4. Digital literacy and access to a smartphone, tablet or computer with internet connection.
5. Continuity in the same workplace for at least 6 months (6) signing the informed consent to participate in the study.

Exclusion Criteria:

1. Diagnosis of serious mental illness.
2. Suicidal ideation.
3. Substance abuse or related disorders.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Intervention Measure (FIM) | Post-treatment 10 weeks from baseline
  Includes 4 items designed to measure appropriateness of the intervention. The scale presents 5-point Likert-type scale (1 = completely disagree, 2 = in disagreement, 3 = neither agree nor disagree, 4 = agree and 5 = completely agree). A total score, ranging from 0 to 20, is calculated by totalling the scores from all the items, and higher total values indicate higher level of Feasibility of the intervention
System Usability Scale (SUS) | Post-treatment, 10 weeks from baseline
  It is a 10-item questionnaire to measure the usability which qualitatively is related with the quality and acceptability of the intervention. The scale presents 5-point Likert-type scale (0 = never, 1 = almost never, 2 = often, 3 = sometimes and 4 = always). A total score, ranging from 0 to 40, is calculated by totalling the scores from all the items, and higher total values indicate higher level of acceptability of the intervention
Client Satisfaction Questionnaire adapted to Internet-Based interventions (CSQ-I) | Post-treatment 10 weeks from baseline
  It is an 8-item, 4-point Likert scale questionnaire that assesses the general satisfaction of the participants regarding the received intervention. The total score ranges from 8 to 32.

SECONDARY OUTCOMES:
Perceived Stress Scale (PSS) | Baseline
  Consists of 10 items in which participants are asked to rate how unpredictable, uncontrollable, and overloaded they have found their life over the past month on a 5-point Likert-type scale. Scores range from 0 to 40, and higher scores reflect higher levels of perceived stress.
Perceived Stress Scale (PSS) | Post-treatment 10 weeks from baseline
  Consists of 10 items in which participants are asked to rate how unpredictable, uncontrollable, and overloaded they have found their life over the past month on a 5-point Likert-type scale. Scores range from 0 to 40, and higher scores reflect higher levels of perceived stress.
Patient Health Questionnaire (PHQ-9) | Baseline
  It is a 9-item scale aimed at screening for depression in primary care and other medical settings. It assesses the frequency of depressive symptoms during the last 2 weeks using a scale from 0 (not at all) to 3 (nearly every day). The total score ranges from 0 to 27, with higher scores indicating higher severity of depression.
Patient Health Questionnaire (PHQ-9) | Post-treatment 10 weeks from baseline
  It is a 9-item scale aimed at screening for depression in primary care and other medical settings. It assesses the frequency of depressive symptoms during the last 2 weeks using a scale from 0 (not at all) to 3 (nearly every day). The total score ranges from 0 to 27, with higher scores indicating higher severity of depression.
General Anxiety Disorder-7 (GAD-7) | Baseline
  It is a 7-item self-reported measure to assess the intensity of anxiety symptoms. It refers to the period of the past 2 weeks; each item is scored in a 4-point Likert-type scale, resulting in a total score that can range from 0 to 21, with higher values reflecting more severe anxiety symptoms.
General Anxiety Disorder-7 (GAD-7) | Post-treatment 10 weeks from baseline
  It is a 7-item self-reported measure to assess the intensity of anxiety symptoms. It refers to the period of the past 2 weeks; each item is scored in a 4-point Likert-type scale, resulting in a total score that can range from 0 to 21, with higher values reflecting more severe anxiety symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Gloria Margarita Guerrero Pertíñez, PhD, Principal Investigator — Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud; José Guzmán Parra, PhD, Principal Investigator — Hospital Regional Universitario de Málaga Plaza del Hospital Civil s/n, Pabellón 4, 1ª Planta, 29009, Málaga
Locations (1):
- Hospital Regional Universitario de Málaga Plaza del Hospital Civil s/n, Pabellón 4, 1ª Planta, 29009, Málaga, Málaga, Spain

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to ethical and privacy considerations. The data collected are sensitive mental health measures from healthcare professionals, and the protocol does not include consent for sharing individual-level data with external researchers. Only aggregated results will be made publicly available.

REFERENCES:
- [Result] Lopez-Del-Hoyo Y, Fernandez-Martinez S, Perez-Aranda A, Monreal-Bartolome A, Barcelo-Soler A, Camarero-Grados L, Armas-Landaeta C, Guzman-Parra J, Carbonell V, Campos D, Chen X, Garcia-Campayo J. Effectiveness of a Web-Based Self-Guided Intervention (MINDxYOU) for Reducing Stress and Promoting Mental Health Among Health Professionals: Results From a Stepped-Wedge Cluster Randomized Trial. J Med Internet Res. 2025 Feb 3;27:e59653. doi: 10.2196/59653. PMID 39899345
- [Result] Lopez-Del-Hoyo Y, Fernandez-Martinez S, Perez-Aranda A, Barcelo-Soler A, Guzman-Parra J, Varela-Moreno E, Campos D, Monreal-Bartolome A, Beltran-Ruiz M, Moreno-Kustner B, Mayoral-Cleries F, Garcia-Campayo J. Effectiveness and implementation of an online intervention (MINDxYOU) for reducing stress and promote mental health among healthcare workers in Spain: a study protocol for a stepped-wedge cluster randomized trial. BMC Nurs. 2022 Nov 10;21(1):308. doi: 10.1186/s12912-022-01089-5. PMID 36357881
- See also: Related Info — https://mindxyou.es/

DOCUMENTS (1):
  • Study Protocol (2025-05-29): https://cdn.clinicaltrials.gov/large-docs/43/NCT07066943/Prot_000.pdf